CLINICAL TRIAL: NCT03346824
Title: Levosimendan Efficacy for Veno-arterial ECMO Weaning: a Retrospective Study
Acronym: LEVO-ECMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6946
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2017-11

CONDITIONS: Cardiogenic Shock
Keywords: Levosimendan; Veno-arterial ECMO; Weaning
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Failure of Weaning from ECMO is a serious complication, reaching an incidence between 29 and 58%. Inotrops are frequently used to help separating patient from ECMO. Levosimendan is an ino-dilatatory medication and was used in different clinical settings. The aim of this study was to evaluate the benefit with levosimendan when used in weaning process.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Patient requiring the need for short-term assistance
* Patient who has agreed to use his medical data for research purposes

Exclusion Criteria:

* Refusal to participate in the study
* Non-weaning attempts due to a death under assistance or a relay by a long-term assistance or heart transplant
* Non-cardiac indications of assistance (indication of pulmonary replacement)
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient who required the use of short-term assistance
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the incidence of weaning failure between patients with levosimendan and others | Data were recorded from admission until 48 hours after weaning from ECMO

CONTACTS AND LOCATIONS:
Locations (1):
- Service Réanimation chirurgicale cardiovasculaire-NHC, Strasbourg, France